CLINICAL TRIAL: NCT07004465
Title: Effectiveness of Vitamin b12 Versus Kenalog in Orabase on Traumatic Ulcer Associated With Orthodontic Treatment: Randomized Control Trial
Brief Title: Effectiveness of Vitamin b12 Versus Kenalog on Traumatic Ulcer Associated With Orthodontic Treatment
Acronym: B12-KEN-TRAUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawraa Ali Abdullah (Other)
Responsible Party: Sponsor-Investigator, Hawraa Ali Abdullah, assist lecturer, Karbala University
Organization: Karbala University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dent/UO-Kerbala/3-14122024; Dent/UO-Kerbala/3-14122024 (Other: kerbala university)
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-06

CONDITIONS: Mouth Ulcer
MeSH Terms: conditions — Oral Ulcer | interventions — Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- vitamin B12 (Experimental): Vitamin B12, also known as cobalamin, is a water-soluble vitamin involved in metabolism
  Interventions: Dietary Supplement: cyanocobalamin
- Kenalog in Orabase (Experimental): The active substance is triamcinolone acetonide 40 mg/ml. The other ingredients are; benzyl alcohol, polysorbate 80, carmellose sodium, sodium chloride and water
  Interventions: Device: triamcinolone acetonide

INTERVENTIONS:
Dietary Supplement: cyanocobalamin — Group A will be given vitamin B12 tablets (1000 mcg) once daily.
  Arms: vitamin B12
Device: triamcinolone acetonide — Group B will be given Kenalog gel (triamcinolone acetonide 40 mg/ml). The other ingredients are benzyl alcohol, polysorbate 80, carmellose sodium, sodium chloride and water, by covering the area twice daily
  Arms: Kenalog in Orabase

SUMMARY:
The study is a randomized controlled trial. the participants will be equally divided into two groups to compare the clinical effectiveness of vitamin b12 versus kenalog in treatment of traumatic ulcers associated with orthodontic treatment during

DETAILED DESCRIPTION:
Recurrent aphthous stomatitis (RAS), commonly called "canker sores," is a perplexing oral condition characterized by the recurrent development of painful aphthous ulcers on non-keratinized oral mucous membranes. Recurrent aphthous stomatitis is a relatively common condition, affecting up to 25% of the worldwide population. Certain factors predispose to RAS, including local trauma, stress, smoking cessation, anemia, and hematinic deficiency. In the patient who undergoes orthodontic management, there is improvement in the dental and facial aesthetics and development of self-confidence. Data also supports the prevalence of traumatic ulcers in the oral cavity and periodontal diseases. Ulcerations can happen due to brackets, bands, arch wires and long unsupported stretches of wire resting against the lips.

Vitamin B12, also known as Cobalamin, is a water-soluble vitamin primarily found in animal products; plays a vital role in the formation of hematopoietic stem cells and vitaminB12 deficiency may play a role in the pathogenesis of recurring aphthous (RAS). TRIAMCINOLONE (Kenalog in Orabase) treats and relieves discomfort caused by mouth sores. It works by decreasing inflammation in the mouth. It belongs to a group of medications called topical steroids.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic adult patients older than 18 years.
* Ulcer due to trauma not more than 10 mm in size.

Exclusion Criteria:

* Patients who had known systemic diseases.
* Concurrent with lesions in the mouth (Bechet's disease, rheumatoid. arthritis, lupus, and acquired immune deficiency syndrome).
* A patient who had received other concurrent treatment for aphthous ulcers.
* Patients with chronic diseases such as liver diseases, rheumatoid arthritis, diabetes, cancer, and renal diseases.
* Pregnant or nursing women.
* Patient who had a known vitamin B12 deficiency.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
pain reduction | 8 days
  The primary outcome will be the reduction in pain intensity at day 4 and day 8 after treatment using a visual analog scale and recording measurements, respectively, for both groups.
  visual analogue scale from 0 cm (no pain) to 10 cm (severe to worst pain), which represents the intensity of subjective experience

SECONDARY OUTCOMES:
ulcer size | 8 days
  measuring ulcer size using vernier will be done on fourth and eighth days for both groups

CONTACTS AND LOCATIONS:
Locations (2):
- Iraq (2):
  - Karbala university, Karbala, Karbala Governorate
  - Kerbala University, Karbala, Kerbala

IPD SHARING:
Plan to Share IPD: No
for ethical consideration

REFERENCES:
- See also: college of dentistry / kerbala university — https://dentistry.uokerbala.edu.iq